CLINICAL TRIAL: NCT03516201
Title: Oral Health in Bariatric Patients
Status: Completed | Type: Observational
Sponsor: University of Göttingen (Other)
Responsible Party: Principal Investigator, Philipp Kanzow, Prof. Dr. med. dent., Dr. rer. medic., Postdoctoral Research Fellow, University of Göttingen
Other Study IDs: 28/3/17
Record Dates: First submitted 2018-03-21; First posted 2018-05-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Adiposity; Dental Diseases; Bariatric Surgery Candidate
Keywords: bariatric surgery; Periodontitis; Caries; erosive tooth wear; Gingivitis; BMI; oral health; obesity
MeSH Terms: conditions — Obesity; Stomatognathic Diseases; Periodontitis; Gingivitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- obese patients after bariatric surgery: obese adults (≥ 18 years) who underwent bariatric surgery
- obese adultes without bariatric surgery: obese adults (≥ 18 years) who did not underwent bariatric surgery at the time of the examination

SUMMARY:
As few is known about the oral health of bariatric patients, this study aimed to analyze the prevalence and severity of erosive tooth wear, dental caries and periodontal diseases of obese patients who underwent bariatric surgery in comparison to obese patients without bariatric procedures.

DETAILED DESCRIPTION:
The prevalence of overweight and obesity is increasing since the 1980s. Being associated with several risk factors such as hypertension, hyperinsulinemia and hyperlipidemia, obesity presents an immediate and long-term health risk for diabetes mellitus, heart diseases, osteoarthritis and certain forms of cancer. For the control of obesity several therapy options have been developed: Beside conservative treatments including change of diet and lifestyle, bariatric surgery is considered as a promising option for patients with severe obesity (BMI ≥ 40 kg/m2). Allowing impressive weight loss from 40 to 80% and effective reduction of comorbidities, bariatric surgery shows some negative/adverse effects as well, like kidney problems, hyperparathyroidism, anemia and metabolic bone diseases. For oral health, two facts are particularly important to consider: Firstly, chronic regurgitation reaching the oral cavity is an important risk factor for erosive tooth wear which initially appear as smooth silky-shining glazed surfaces. Further progress is often associated with hypersensitivities and aesthetic deficits. Over time, often substantial loss can been observed, provoking hypersensitivities and aesthetic deficits. Secondly, depending on the type of bariatric surgery, pronounced postoperative metabolic and nutritional changes can be observed which also might influence oral health. Aim of this study is to analyze the prevalence and severity of erosive tooth wear, dental caries and periodontal diseases of obese patients who underwent bariatric surgery in comparison to obese patients without bariatric procedures.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* BMI ≥ 25 kg/m2 without or after bariatric surgery

Exclusion Criteria:

* refusal for participation
* age <18 years
* BMI <25 kg/m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study enrolls obese adults (Age over 18 years) with an BMI (body mass index) of at least 25 kg/m2 without or after bariatric surgery
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2018-06-15 (Actual); Primary Completion 2020-02-12 (Actual); Study Completion 2020-02-12 (Actual)

PRIMARY OUTCOMES:
Oral health of obese adults without bariatric surgery - attachment loss | 10-15 Minutes
  probing depths (mm) + recessions (mm)
Oral health of obese adults without bariatric surgery - BOP | 2 Minutes
  BOP (Bleeding on probing, %) as indicator of inflammation
Oral health of obese adults without bariatric surgery - dental caries | 2-5 Minutes
  ICDAS (International Caries Detection and Assessment System II, 0-6), presence of restaurations/ crowns (yes/no): calculation of DMFT
Oral health of obese adults without bariatric surgery - erosive tooth wear | 1-2 Minutes
  BEWE (Basic erosive wear examination, 0-3)

SECONDARY OUTCOMES:
Oral health of obese adults after bariatric surgery - attachment loss | 10-15 Min
  probing depths (mm) + recessions (mm)
Oral health of obese adults after bariatric surgery - BOP | 2 Minutes
  BOP (Bleeding on probing, %) as indicator of inflammation
Oral health of obese adults after bariatric surgery - dental caries | 2-5 Minutes
  ICDAS (International Caries Detection and Assessment System II, 0-6), presence of restaurations/ crowns (yes/no): calculation of DMFT
Oral health of obese adults after bariatric surgery - erosive tooth wear | 1-2 Minutes
  BEWE (Basic erosive wear examination, 0-3)

CONTACTS AND LOCATIONS:
Overall Officials: Annette Wiegand, Prof. Dr. med. dent., Study Director — Dept. of Prev. Dentistry, Periodontology and Cariology
Locations (1):
- Dept. of Prev. Dentistry, Periodontology and Cariology, University Medical Center Göttingen, Göttingen, Germany